CLINICAL TRIAL: NCT00757614
Title: A Population Based Study of Genetic Predisposition and Gene-Environment Interactions in Cancer in East Anglia, Trent and West Midlands
Brief Title: Study of Genes and Environment in Patients With Cancer in East Anglia, Trent, or West Midlands Regions of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598879; MREC-SEARCH-CANCER; MREC-07/MRE05/17
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2010-04

CONDITIONS: Bladder Cancer; Brain and Central Nervous System Tumors; Esophageal Cancer; Intraocular Melanoma; Kidney Cancer; Lymphoma; Melanoma (Skin); Pancreatic Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: AIDS-related lymphoma; cutaneous lymphoma; adult Hodgkin lymphoma; adult non-Hodgkin lymphoma; intraocular lymphoma; adult T-cell leukemia/lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; noncutaneous extranodal lymphoma; adult astrocytic tumors; adult brain stem glioma; adult choroid plexus tumor; adult craniopharyngioma; adult embryonal tumor; adult ependymal tumors; adult meningeal tumor; adult oligodendroglial tumors; adult pineal parenchymal tumor; adult brain tumor; intraocular melanoma; bladder cancer; clear cell sarcoma of the kidney; congenital mesoblastic nephroma; esophageal cancer; melanoma; pancreatic cancer; peripheral primitive neuroectodermal tumor of the kidney; renal cell carcinoma; rhabdoid tumor of the kidney; transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Central Nervous System Neoplasms; Esophageal Neoplasms; Uveal Melanoma; Kidney Neoplasms; Lymphoma; Melanoma; Pancreatic Neoplasms; Lymphoma, AIDS-Related; Lymphoma, T-Cell, Cutaneous; Hodgkin Disease; Lymphoma, Non-Hodgkin; Intraocular Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Astrocytoma; Choroid Plexus Neoplasms; Craniopharyngioma; Neoplasms, Germ Cell and Embryonal; Meningeal Neoplasms; Pinealoma; Brain Neoplasms; Nephroma, Mesoblastic; Carcinoma, Renal Cell | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: DNA analysis
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility to cancer and interactions between genes and the environment in patients with cancer in East Anglia, Trent, or West Midlands of the United Kingdom.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain epidemiological information and biological material on a population-based series of cancer cases, including malignant melanoma, lymphoma, bladder, kidney, esophageal, and pancreatic cancer, and brain tumors.
* Identify novel cancer susceptibility genes, by comparison of genotype frequencies in cases with the corresponding frequencies in large control series.
* To estimate the age and sex-specific risks associated with variants in predisposition genes.
* To evaluate interactions between polymorphisms in predisposition genes and potential lifestyle risk factors.

OUTLINE: This is a multicenter study.

Patients complete a detailed epidemiological questionnaire that includes information on education, occupation, smoking habits, alcohol consumption, height, weight, reproductive history (age at menarche, age at pregnancies, parity, and age at menopause), oral contraceptive use, hormone replacement therapy use, family history of cancer, and past medical history.

Blood samples are collected from patients. DNA is extracted from these blood samples, from samples collected from cancer-free control participants in MREC-SEARCH-CONTROL, and from additional controls through the European Prospective Investigation of Cancer (EPIC) study (a population-based study of diet and health based in Norfolk, East Anglia). DNA samples are analyzed for polymorphisms of low penetrance cancer susceptibility genes.

In addition to the cancer patients recruited for this study, patients with breast, ovarian, endometrial, colorectal, and prostate cancer are recruited for the following related clinical trials: MREC-SEARCH-BREAST, MREC-SEARCH-OVARIAN, MREC-SEARCH-ENDOMETRIAL, MREC-SEARCH-COLORECTAL, and MREC-SEARCH-PROSTATE.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosed with bladder cancer, kidney cancer, esophageal cancer, pancreatic cancer, brain cancer, malignant melanoma, or lymphoma within the past 5 years
* Identified through the Cancer Research Network OR through the cancer registry serving any of the following geographic regions of the United Kingdom:

  * East Anglia
  * West Midlands
  * Trent

PATIENT CHARACTERISTICS:

* Identified by the patient's general practitioner as fit to contact for this study
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of epidemiological information and biological material
Identification of novel cancer susceptibility genes
Estimation of the age and sex-specific risks associated with variants in predisposition genes
Evaluation of interactions between polymorphisms in predisposition genes and potential lifestyle risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom